CLINICAL TRIAL: NCT00346996
Title: The Effect of Insulin Analogues and Human Insulin on the Incidence of Severe Hypoglycaemia in Hypoglycaemia Prone Type 1 Diabetic Patients
Brief Title: Insulin Analogues and Severe Hypoglycaemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lise Tarnow (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor-Investigator, Lise Tarnow, professor, Steno Diabetes Center Copenhagen
Organization: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HypoAna
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Type 1 Diabetes
Keywords: diabetes; insulin; insulin analogues; hypoglycaemia; severe hypoglycaemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance; Hypoglycemia | interventions — Insulin Aspart; Isophane Insulin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): HUman Insulin
  Interventions: Drug: human insulin /insulin isophane
- 2 (Experimental): Analogue insulin
  Interventions: Drug: insulin levemir / aspart

INTERVENTIONS:
Drug: insulin levemir / aspart — for subcutaneous injection
  Arms: 2
Drug: human insulin /insulin isophane — for subcutaneous injection
  Arms: 1

SUMMARY:
Severe hypoglycaemia is hampering the lives of many diabetic patients. The effect on the occurrence of severe hypoglycaemia during two different insulin regimens are to be investigated. In total, 250 hypoglycaemia prone type 1 diabetic patients will be randomised to receive analogue and human insulin for one year in random order. Outcomes will be number of episodes of severe hypoglycaemia

DETAILED DESCRIPTION:
The primary objective is to evaluate the effects of insulin analogue and human insulin on incidence of severe hypoglycaemia in type 1 diabetic patients prone to hypoglycaemia.Secondary endpoints are effect on incidence of symptomatic and asymptomatic documented hypoglycaemia.

Study Design: An open, randomised, controlled, cross-over multi-centre study. Each treatment period lasts for one year. Patients will be randomised to treatment with basal bolus therapy with insulin detemir / aspart and insulatard / actrapid in random order. Endpoints will be assessed during the last 9 months of each treatment arm.

Patient population: 250 type 1 diabetic patients with a history of two or more episodes of severe hypoglycaemia during the preceding year.

Interventions: Basal bolus therapy with insulin detemir / aspart and insulatard / human actrapid in random order. Each treatment period lasts 12 months.

Methods: Patients will record all events of severe hypoglycaemia, documented symptomatic and asymptomatic hypoglycaemia in a diary and report all events of severe hypoglycaemia by telephone within 24 hours. All patients will be instructed to do and record home blood glucose monitoring (SMBG) i.e. 7 point profiles twice per week and nocturnal measurements once every month.

Outcomes: Severe hypoglycaemia, documented symptomatic and asymptomatic hypoglycaemia Efficacy: Number of reported episodes of severe, documented symptomatic and asymptomatic hypoglycaemia during the last 9 months of treatment - during daytime and night time.

Safety: Adverse reactions

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for 5 years.
* Age>18 years.
* Two or more episodes of hypoglycaemia during the last year,

Exclusion Criteria:

* History of Addisons disease
* Growth hormone deficiency or untreated myxoedema
* CVD within 6 months
* Cancer within 5 years
* Alcohol or drug abuse
* Pregnant or lactating women
* Fertile women without effective contraception
* Participation in another trial within 30 days
* Inability to understand the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2007-05; Primary Completion 2011-11 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Severe hypoglycaemia | 9 months

SECONDARY OUTCOMES:
asymptomatic hypoglycaemia | 9 months
hypoglycaemia during nighttime | 9 months
hypoglycaemia during daytime | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Lise Tarnow, MD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Denmark

REFERENCES:
- [Derived] Pedersen-Bjergaard U, Kristensen PL, Norgaard K, Perrild H, Jensen T, Thorsteinsson B, Nikolajsen A, Tarnow L. Short-term cost-effectiveness of insulin detemir and insulin aspart in people with type 1 diabetes who are prone to recurrent severe hypoglycemia. Curr Med Res Opin. 2016 Oct;32(10):1719-1725. doi: 10.1080/03007995.2016.1205006. Epub 2016 Jul 20. PMID 27326862
- [Derived] Agesen RM, Kristensen PL, Beck-Nielsen H, Norgaard K, Perrild H, Christiansen JS, Jensen T, Hougaard P, Parving HH, Thorsteinsson B, Tarnow L, Pedersen-Bjergaard U. Effect of insulin analogues on frequency of non-severe hypoglycaemia in patients with type 1 diabetes prone to severe hypoglycaemia: The HypoAna trial. Diabetes Metab. 2016 Sep;42(4):249-55. doi: 10.1016/j.diabet.2016.03.001. Epub 2016 Apr 7. PMID 27068361
- [Derived] Pedersen-Bjergaard U, Kristensen PL, Beck-Nielsen H, Norgaard K, Perrild H, Christiansen JS, Jensen T, Hougaard P, Parving HH, Thorsteinsson B, Tarnow L. Effect of insulin analogues on risk of severe hypoglycaemia in patients with type 1 diabetes prone to recurrent severe hypoglycaemia (HypoAna trial): a prospective, randomised, open-label, blinded-endpoint crossover trial. Lancet Diabetes Endocrinol. 2014 Jul;2(7):553-61. doi: 10.1016/S2213-8587(14)70073-7. Epub 2014 May 2. PMID 24794703
- [Derived] Kristensen PL, Pedersen-Bjergaard U, Beck-Nielsen H, Norgaard K, Perrild H, Christiansen JS, Jensen T, Parving HH, Thorsteinsson B, Tarnow L. A prospective randomised cross-over study of the effect of insulin analogues and human insulin on the frequency of severe hypoglycaemia in patients with type 1 diabetes and recurrent hypoglycaemia (the HypoAna trial): study rationale and design. BMC Endocr Disord. 2012 Jun 22;12:10. doi: 10.1186/1472-6823-12-10. PMID 22727048